CLINICAL TRIAL: NCT05870384
Title: Effects of Group Interpersonal Psychotherapy (IPT-G) Applied to Family Members Who Caregivers of Patients With Schizophrenia on Caregiver Burden, Social Support, Expression of Emotion, Stigma, and Adherence to Treatment
Brief Title: Application of Group Interpersonal Psychotherapy (IPT-G) to Family Members Caring for Patients With Schizophrenia
Acronym: IPT-G
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: People didn't apply. The number of participants required to begin the intervention was not reached.
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Melisa BULUT, Research Assistant, Abant Izzet Baysal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AIBU-PSK-MB-01
Record Dates: First submitted 2023-03-25; First posted 2023-05-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Interpersonal Psychotherapy; Family Caregivers
Keywords: Interpersonal Psychotherapy; Schizophrenia; Caregiver Burden; Social Support; Social Stigma; Treatment Adherence and Compliance; Expressed Emotion
MeSH Terms: conditions — Schizophrenia; Caregiver Burden; Social Stigma; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This study is a single group Remeasurement Quasi-experimental Study. The intervention in the study is the application of IPT-G to the caregivers of the patients with schizophrenia. The intervention consists of 10 sessions to be held once a week. The first 2 sessions will be individual, followed by 8 group sessions. Sessions will last an average of 90 minutes. The group is a closed group, no new participants will be accepted after the sessions have started. The study will measure the impact of the therapy on both the caregivers and patients, with follow-up evaluations at 3 and 6 months after the sessions. At the end of the experiment, the "t-test for dependent groups" will be used, in which the averages of the pre-test and post-test scores are compared whether the results are significant or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychotherapy (Experimental): Group psychotherapy will be applied to a single intervention group.
  Interventions: Behavioral: Group Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Group Interpersonal Psychotherapy — Ten sessions of IPT-G, which focuses on the common problem area of patient relatives, will be applied.

SUMMARY:
The goal of this re-measured quasi-experimental study is to evaluate the effect of Group Interpersonal Psychotherapy (IPT-G) intervention given to caregiver family members of people with schizophrenia on caregiver burden, perception of social support and stigma, adherence to treatment in people with schizophrenia they care for, and emotional expression in both caregivers and people with schizophrenia they care for. The main hypotheses it aims to test are:

1. IPT-G intervention will reduce the caregiver burden of caregivers of individuals with schizophrenia.
2. IPT-G intervention will increase the perceived social support levels of caregivers of individuals with schizophrenia.
3. IPT-G intervention will reduce the level of stigma of caregivers of individuals with schizophrenia.
4. IPT-G intervention will reduce the level of emotional expression of caregivers of individuals with schizophrenia.
5. IPT-G intervention applied to caregivers will increase the level of adherence to treatment of individuals with schizophrenia they care for.
6. IPT-G intervention applied to caregivers will reduce the emotional expression levels of individuals with schizophrenia they care for.

DETAILED DESCRIPTION:
Family members who care for individuals with a chronic mental illness such as schizophrenia are exposed to many risks such as stress, fatigue, depression, care burden, stigma, problems in family and interpersonal relationships, conflicts, financial difficulties, social isolation, disruption of daily routines. IPT is a short-term psychotherapy that works on specific interpersonal problem areas associated with depression, anxiety, and general psychological distress. IPT focuses on the following interpersonal problem areas: grief or complicated dispute, bereavement, role, role transition, interpersonal deficits . In these problem areas, IPT is applied individually as well as as group psychotherapy. IPT-G is carried out with group members who share a common distress. IPT-G is more structured than individual IPT. There is a practitioner's guide. IPT-G has a specific agenda, structure and defined endpoint. In IPT-G, the group usually has 6-10 members. Sessions last approximately 90 minutes. The main objectives of IPT-G can be summarized as 1) psychoeducation, 2) increasing social support, 3) solving interpersonal problems. In this sense, the application of IPT-G in the caregivers of individuals with schizophrenia may be promising both for the caregivers and the patients they care for. Therefore, family members who care for individuals diagnosed with schizophrenia living in Turkey/Bolu province, who are willing to participate in the IPT-G intervention, and who meet the inclusion/exclusion criteria of the study will constitute the sample of the study. Participants will be selected from the caregivers of the patients reached from Bolu Abant İzzet Baysal University, İzzet Baysal Training and Research Hospital and Bolu İzzet Baysal Mental Health and Diseases Hospital. A poster inviting the caregivers of the patients will be prepared and hung in the hospitals. Group psychotherapy intervention for the caregivers of patients who meet the inclusion and exclusion criteria of the study will be carried out in a training room in Bolu Abant İzzet Baysal University, Faculty of Health Sciences, Department of Nursing, where the researchers work. The group therapy will be made by the researcher, a licensed psychotherapist. IPT-G will only be applied to caregivers. No application will be made to the patients. In addition, it will be measured whether the intervention applied to the caregivers indirectly has any effect on the patient. Persons to be included in the application will be informed about the application. Signed consent will be obtained. In order to include individuals in the IPT-G intervention, the researcher who will conduct the application will conduct two one-on-one interviews with caregivers to evaluate whether they are suitable for group intervention. The therapist will include caregivers with a similar problem focus in the group. Since it is suggested that the IPT-G group intervention should consist of 6-10 people, this number will be taken as the basis. Group therapy will be done once a week. Sessions will last approximately 90 minutes. The intervention will be completed in a total of ten sessions, with two-session individual interviews and eight-session group sessions. Measurement tools will be applied to caregivers and the patients they care for at the beginning of the group therapy, at the end of the last session, at the end of the third month following the end of the sessions, and at the end of the sixth month following the end of the sessions. A total of four measurements will be made. Scales and sociodemographic data form will be used as data collection tools.Sociodemographic data collection form, Emotional Expression Scale Caregiver Version, Stigma Scale for the Families of Psychiatric Patients (SCFPP), Zarit Caregiver Burden Interview, Multidimensional Scale of Perceived Social Support will be administered face-to-face to caregivers in the IPT-G intervention. The Patient Version of the Emotion Expression Scale and The Medication Adherence Report Scale will be applied to the individuals diagnosed with schizophrenia, who are cared for by the caregivers in the IPT-G intervention.At the end of the experiment, the "t-test for dependent groups" will be used, in which the averages of the pre-test and post-test scores are compared whether the results are significant or not.The research complies with the ethical principles of benefit and non-harm. There is no aspect of the research that could pose a risk or cause harm to the participants. The research intervention is envisaged to provide beneficial outcomes to the participants. Shares made during individual interviews and group sessions will be kept confidential under the principle of protecting privacy. Privacy and confidentiality is the norm of the group and compliance by all participants will be contractually assured and encouraged. Researchers will not share therapy notes unless they pose a risk to the individual, his/her environment and other third parties, unless there is a judicial process.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65
* Being able to speak and understand fluent Turkish,
* Being the primary caregiver of a family member with one of the Schizophrenic Disorders and Psychotic Disorders,
* Caring for a family member with Schizophrenia and Schizophrenia Spectrum Disorder for at least 6 months.
* Both the caregiver and the patient voluntarily agree to participate in the study.

Exclusion Criteria:

* Having a dismissive attachment style (to be evaluated by the researcher),
* Having antisocial personality traits (to be evaluated by the researcher),
* Having narcissistic personality traits (to be evaluated by the researcher),
* Having active suicidal ideation (to be evaluated by the investigator).

Removal criteria:

* Not attending more than two sessions of the 7-session intensive/group phase
* Failure to comply with the norms and rules of group therapy (continuity, confidentiality, respectful communication, interaction with group members, participation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver burden evaluated with the Zarit Caregiver Burden Scale (ZCBS) | Change in caregiver burden at 6 months
  The primary outcome measure of the study is the care burden. Caregivers' burden will be evaluated with repeated tests before and after the intervention. For this, the "Zarit Caregiver Burden Scale (ZCBS)" scale will be used.The scale will be applied only to caregivers who participate in the group psychotherapy intervention.
  Zarit Caregiver Burden Scale (ZCBS): The scale consists of 22 items. It includes the negative effects of caregiving on physical, mental health, social activity and economic resources.The total score varies between 22-110. The higher the scores, the higher the level of burden. It is expected that the burden of care score will decrease in the measurements made after the intervention.

SECONDARY OUTCOMES:
Change in expression of emotion evaluated with Expression of Emotion Scale and Level of Expressed Emotion Scale | Change in expression of emotion at 6 months
  Expression of emotion will be measured both in caregivers participating in group psychotherapy intervention and in patients they care for without intervention with repeated tests before and after the intervention.
  Expression of Emotion Scale: This scale will be filled by caregivers. The scale consists of 41 "true/false" questions. The higher the scores, the higher the level of emotional expression. The total score ranges from 0 to 41.It is expected that the expression of emotion score will decrease in the measurements made after the intervention.
  Level of Expressed Emotion Scale:This scale will be filled by patients. The scale asks patients to evaluate the attitude of their caregivers towards them. The scale consists of 60 "true/false" questions. The total score ranges from 0 to 60.It is expected that the expression of emotion score will decrease in the measurements made after the intervention.
Change in stigma evaluated with the Stigma Scale for the Families of Psychiatric Patients (SCFPP) | Change in stigma at 6 months
  Stigma will be evaluated with repeated tests before and after the intervention. For this, the "Stigma Scale for the Families of Psychiatric Patients (SCFPP)" scale will be used.The scale will be applied only to caregivers who participate in the group psychotherapy intervention.
  Stigma Scale for the Families of Psychiatric Patients (SCFPP): The scale consists of 17 items. Scoring of the scale is made as the lowest 1 and the highest 3 points; cut-off score was calculated as 1.67.The higher the scores, the higher the level of stigma.It is expected that the stigma score will decrease in the measurements made after the intervention.
Change in perceived social support evaluated with the Multidimensional Scale of Perceived Social Support (MSPSS) | Change in perceived social support at 6 months
  Perceived social support will be evaluated with repeated tests before and after the intervention. For this, the "Multidimensional Scale of Perceived Social Support (MSPSS)" scale will be used.The scale will be applied only to caregivers who participate in the group psychotherapy intervention.
  Multidimensional Scale of Perceived Social Support (MSPSS): The scale consists of 12 items. The total score varies between 0-84. A high score indicates high perceived social support. It is expected that the perceived social support score will increase in the measurements made after the intervention.
Change in medication adherence evaluated with the Medication Adherence Rating Scale (MARS) | Change in medication adherence at 6 months
  Medication adherence will be evaluated with repeated tests before and after the intervention. For this, the "Medication Adherence Rating Scale (MARS)" scale will be used.The scale will be applied to patients cared for by caregivers participating in the intervention.
  Medication Adherence Rating Scale (MARS):The scale consists of 10 "yes/no" questions.The total score varies between 1-10.Low scores on the scale indicate poor adherence to treatment, and high scores indicate high adherence to treatment. 1 and 7 points shows that poor adherence to treatment, between 8 and 10 were high. It is expected that the perceived social support score will increase in the measurements made after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Bulut, Study Director — Bolu Abant İzzet Baysal University; Nazmiye Yıldırım, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Faculty of Health Sciences, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuijpers P, Donker T, Weissman MM, Ravitz P, Cristea IA. Interpersonal Psychotherapy for Mental Health Problems: A Comprehensive Meta-Analysis. Am J Psychiatry. 2016 Jul 1;173(7):680-7. doi: 10.1176/appi.ajp.2015.15091141. Epub 2016 Apr 1. PMID 27032627
- [Background] Arslantas H. The burden of schizophrenia on caregivers. Current Approaches in Psychiatry. 2011; 3(2):251-277.
- [Background] Chang KH, Horrocks S. Lived experiences of family caregivers of mentally ill relatives. J Adv Nurs. 2006 Feb;53(4):435-43. doi: 10.1111/j.1365-2648.2006.03732.x. PMID 16448486
- [Background] Stuart S, Schultz J. IPT for Groups Clinician's Handbook. IPT Institute. 2016
- [Background] Chen WY, Lukens E. Well being, depressive symptoms, and burden among parent and sibling caregivers of persons with severe and persistent mental illness. Social Work in Mental Health. 2011; 9(6): 397-416.
- [Result] Durmaz H, Okanli A. Effects of interpersonal psychotherapy (ipt) techniques and psychoeducation on self-efficacy and care burden in families of patients with schizophrenia. American Journal of Family Therapy. 2021; 49(4): 373-391.
- [Result] Mutamba BB, Kane JC, de Jong JTVM, Okello J, Musisi S, Kohrt BA. Psychological treatments delivered by community health workers in low-resource government health systems: effectiveness of group interpersonal psychotherapy for caregivers of children affected by nodding syndrome in Uganda. Psychol Med. 2018 Nov;48(15):2573-2583. doi: 10.1017/S0033291718000193. Epub 2018 Feb 15. PMID 29444721
- [Result] Glanville DN, Dixon L. Caregiver burden, family treatment approaches and service use in families of patients with schizophrenia. Isr J Psychiatry Relat Sci. 2005;42(1):15-22. PMID 16134403